CLINICAL TRIAL: NCT03894501
Title: Mindfulness Oriented Recovery Enhancement as an Adjunct to Methadone Treatment for Opioid Use and Chronic Pain Management Pilot
Brief Title: Pilot of Mindfulness Oriented Recovery Enhancement in MethadoneTreatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: University of Utah (Other)
Responsible Party: Principal Investigator, Nina A. Cooperman, Psy. D., Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018001127
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Results first posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-11

CONDITIONS: Opioid Use; Chronic Pain
Keywords: opioid; chronic pain; methadone; mindfulness
MeSH Terms: conditions — Chronic Pain | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Two-arm randomized controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Oriented Recovery Enhancement (Experimental): The Mindfulness Oriented Recovery Enhancement arm will participate in eight, weekly, two-hour group sessions.MORE sessions involve mindfulness training to prevent opioid relapse and reduce pain, cognitive reappraisal to decrease negative affect and regulate opioid craving, and savoring to augment natural reward processing and evoke positive emotion. Each session begins with a mindful breathing meditation, followed by a debriefing session. The therapist then debriefs participants' homework practice of using mindfulness, reappraisal, and savoring skills to cope with pain and enhance well-being in everyday life. During this debrief of the homework. Next, new psychoeducational material is introduced. Sessions culminate with an experiential exercise, and close with a brief mindful breathing meditation. Participants are asked to practice 15 minutes of mindfulness/reappraisal/savoring skills each day.
  Interventions: Behavioral: Mindfulness Oriented Recovery Enhancement
- Methadone program behavioral treatment as usual (Other): In the methadone programs, clients typically come to the clinic regularly to get their methadone dose. Clients see their clinic substance abuse counselor for individual counseling, usually weekly at the beginning of treatment, with decreasing frequency if they remain abstinent and progress through treatment. Depending on clients' stage of MMT and success with remaining abstinent from drugs, they may be required to attend clinic treatment groups. Also, some clients may choose to go to voluntary counseling, educational, or support groups.
  Interventions: Behavioral: Methadone program behavioral treatment as usual

INTERVENTIONS:
Behavioral: Mindfulness Oriented Recovery Enhancement — MORE sessions involve mindfulness training to prevent opioid relapse and reduce pain, cognitive reappraisal to decrease negative affect and regulate opioid craving, and savoring to augment natural reward processing and evoke positive emotion. Each session begins with a mindful breathing meditation, followed by a debriefing session. The therapist then debriefs participants' homework practice of using mindfulness, reappraisal, and savoring skills to cope with pain and enhance well-being in everyday life. During this debrief of the homework. Next, new psychoeducational material is introduced. Sessions culminate with an experiential exercise, and close with a brief mindful breathing meditation. Participants are asked to practice 15 minutes of mindfulness/reappraisal/savoring skills each day.
  Other Names: MORE
  Arms: Mindfulness Oriented Recovery Enhancement
Behavioral: Methadone program behavioral treatment as usual — In the methadone programs, clients typically come to the clinic regularly to get their methadone dose. Clients see their clinic substance abuse counselor for individual counseling, usually weekly at the beginning of treatment, with decreasing frequency if they remain abstinent and progress through treatment. Depending on clients' stage of MMT and success with remaining abstinent from drugs, they may be required to attend clinic treatment groups. Also, some clients may choose to go to voluntary counseling, educational, or support groups.
  Other Names: Treatment as Usual, TAU
  Arms: Methadone program behavioral treatment as usual

SUMMARY:
This pilot study aims to evaluate the impact of a novel intervention, Mindfulness Oriented Recovery Enhancement (MORE), on opioid use and chronic pain among individuals receiving methadone maintenance treatment (MMT). The main goal of this pilot study is to test the feasibility of our study methods before conducting a clinical trial to assess MORE with respect to a range of clinical outcomes. This study will involve a 2-arm individually randomized controlled trial design that compares MORE and treatment as usual (TAU).

DETAILED DESCRIPTION:
This pilot study is a 2-arm individually randomized controlled trial design in which outcomes of MMT patients randomized to MORE are compared to outcomes of those randomized to treatment as usual (TAU). In the pilot study (R21; N=30), we will randomize MMT patients with chronic pain to MORE (n=15) or TAU (n=15). This study phase will focus on establishing study feasibility in recruiting, retaining, and following up study participants before progressing to a larger Phase II clinical trial (R33, N=150). Participants with pain who are receiving MMT for an opioid use disorder (OUD) will be recruited from two methadone clinics in New Jersey.

Participants will be recruited through flyers posted in the clinics, being approached by research assistants in the waiting room of their usual methadone clinic, and referral by clinic staff. The number of individuals who contact the study staff through the flyers or referral and who are approached by study staff in the clinics will be tracked. Number of individuals who refuse study participation and who consent to the study will also be tracked. If an individual is interested in study participation, a trained research assistant will lead the individual through the informed consent process in a private space.

Since MORE is a closed group, we will randomize cohorts of 14-16 participants (depending on speed of recruitment) at each site to TAU or MORE with block randomization. Once we 14-16 participants at a particular clinic, we will randomize participants to MORE or TAU, and the MORE group will begin.

Participants randomized to the MORE condition will participate in eight, weekly, two-hour group sessions led by a clinic or study counselor. Each session will contain 6-8 participants and take place in a private room at the methadone clinic. Attendance at each session and reasons for missing sessions will be recorded Participants randomized to the control condition will continue receiving treatment as usual.

All study participants will partake in a total of three interviews lasting up to 90 minutes and occurring at baseline, 8- and 16- weeks post-baseline in private rooms in the methadone clinics. Each participant will also have a urine or saliva sample collected during each assessment. All attempts to reach participants to schedule follow-up assessments will be tracked. Participants will also complete cognitive testing (for approx. 30-45 minutes) at baseline and 8-weeks and ecological momentary assessments (EMA) conducted via smartphones, which will be provided to each participant by study staff. EMA participation will require the participant to respond to twice-daily prompts in which they will be asked a series of brief questions regarding their current mood and exposure to opioid triggers. Additionally, subjects will be asked to initiate responses when they experience serious craving or relapse to opioid use. Each EMA assessment will last approximately 3-5 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* English-speaking
* Been in methadone treatment for at least 3 months
* Experience a non-malignant pain (with an intensity level of 8 or higher on the Gracely Box Scale) for a duration of 2 months or longer.

Exclusion Criteria:

* Exhibit cognitive impairment (score <24 on the Mini Mental Status Exam)
* Exhibit psychosis (positive SCID Psychotic Screen),
* Are at suicidal risk (positive score on ASQ Suicide Risk Screening Tool)
* Unable to attend group sessions due to distance, work, commitments or other logistical problems,
* Are currently pregnant or breastfeeding
* Are planning to be pregnant or breastfeeding the next 16 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nina A Cooperman, PsyD, Principal Investigator — Rutgers Robert Wood Johnson Medical School
Locations (1):
- Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Analyses of data generated from this project will be shared with the scientific community through publications in peer-reviewed journals and presentations at scientific meetings. The proposed research will include data from approximately 30 individuals in methadone maintenance treatment. The final dataset will include self-reported demographic and behavioral data from interviews with the subjects and laboratory data from urine specimens provided. Because we will be following study participants, we will be collecting identifying information. The final dataset will be stripped of identifiers prior to release for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 36 months after study publication.
Access Criteria: We will make the data and associated documentation available to research community scientists only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- [Result] Garland EL, Hanley AW, Kline A, Cooperman NA. Mindfulness-Oriented Recovery Enhancement reduces opioid craving among individuals with opioid use disorder and chronic pain in medication assisted treatment: Ecological momentary assessments from a stage 1 randomized controlled trial. Drug Alcohol Depend. 2019 Oct 1;203:61-65. doi: 10.1016/j.drugalcdep.2019.07.007. Epub 2019 Aug 5. PMID 31404850

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mindfulness Oriented Recovery Enhancement | Methadone Program Behavioral Treatment as Usual
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness Oriented Recovery Enhancement | Methadone Program Behavioral Treatment as Usual | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (8.7) | 52.9 (8.4) | 50.4 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 7 | 8 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 9 | 16
  White | 7 | 4 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 15
Days of Illicit Drug Use [Mean (Standard Deviation); unit: days] — Research staff asked participants if they used various drugs (i.e., heroin, cocaine, opioids, marijuana, amphetamines, inhalants, hallucinogens, benzodiazepines, zolpidem, methylphenidate, or other drugs) in the past 30 days and the number of days of use for each drug in the past 30 days. "Days of illicit drug use" was determined by counting the number of days each participant used drugs based on past-30 day self-reports at the baseline assessment.
  days | 24.0 (17.4) | 25.2 (29.3) | 24.6 (23.7)
Days of Illicit Opioid Use [Mean (Standard Deviation); unit: days] — Research staff asked participants if they used illicit opioids in the past 30 days and the number of days of use for each drug in the past 30 days. "Days of illicit opioid use" was determined by counting the number of days each participant used illicit opioids based on past-30 day self-reports at the baseline assessment.
  days | 6.4 (9.2) | 11.7 (12.8) | 9.1 (11.3)
Pain Level [Mean (Standard Deviation); unit: score on a scale] — Pain was assess with the pain subscale (i.e., bodily pain severity and interference) of the RAND 36-Item Short Form Health Survey. Scores range from 0 to 100, with higher scores indicating better functioning, health, and well-being and less pain, limitations, and symptom severity or interference as compared to lower scores.
  score on a scale | 28.3 (27.6) | 37.5 (23.5) | 32.9 (25.6)
Depression Level [Mean (Standard Deviation); unit: score on a scale] — Depression was measured with Center for Epidemiologic Studies Depression Scale (CES-D). The CES-D scale is a widely used valid and reliable measure that consists of 20 items with potential scores ranging from 0 to 60. A score above 16 on the CES-D indicates clinically significant symptoms of depression. Higher scores on the CES-D indicates greater depression.
  score on a scale | 27.2 (15.3) | 23.5 (13.4) | 25.4 (14.2)
Anxiety Level. [Mean (Standard Deviation); unit: score on a scale] — Anxiety was measured with the Beck Anxiety Inventory (BAI). The BAI is also a widely used, reliable, and valid scale that consists of 21 items with potential scores ranging from 0 to 63. A score of 16 or higher indicates clinically significant symptoms of anxiety. A higher score on the BAI indicates greater anxiety.
  score on a scale | 41.7 (14.5) | 39.7 (12.3) | 40.7 (13.2)

OUTCOME MEASURES:

1. Primary Outcome: Study Interest
Description: The number of individuals who express interest in the study.
Time Frame: Baseline
Population: Methadone clinic clients.
Measure: Count of Participants; unit: Participants
Groups:
- Participants Who Expressed Interest in the Study: Individuals who asked for information on the study or who asked to be screened for eligibility.
Arm/Group | Participants Who Expressed Interest in the Study
Number analyzed (Participants) | 32
Participants | 32

2. Primary Outcome: Study Refusal
Description: The number of individuals who who refuse participation when offered.
Time Frame: Baseline
Population: Individuals who expressed interest in the study.
Measure: Count of Participants; unit: Participants
Groups:
- The Number of Individuals Who Who Refuse Study Participation When Offered.: The number of individuals who who refuse study participation when offered.
Arm/Group | The Number of Individuals Who Who Refuse Study Participation When Offered.
Number analyzed (Participants) | 32
Participants | 2

3. Primary Outcome: Individuals Screened
Description: The number of individuals screened and eligible/ineligible.
Time Frame: Baseline (study enrollment)
Population: Individuals screened for eligibility.
Measure: Count of Participants; unit: Participants
Groups:
- The Number of Individuals Screened and Ineligible.: The number of individuals screened and ineligible.
Arm/Group | The Number of Individuals Screened and Ineligible.
Number analyzed (Participants) | 32
Participants | 0

4. Primary Outcome: Individuals Consented.
Description: The number of individuals consented.
Time Frame: Baseline (study enrollment)
Population: Eligible individuals.
Measure: Count of Participants; unit: Participants
Groups:
- The Number of Eligible Participants Consented: The number of eligible individuals consented.
Arm/Group | The Number of Eligible Participants Consented
Number analyzed (Participants) | 32
Participants | 31

5. Primary Outcome: Refusal After/During Consent Process.
Description: The number of individuals who refuse participation after/during consent process.
Time Frame: Enrollment
Population: Individuals who participated in consent process.
Measure: Count of Participants; unit: Participants
Groups:
- The Number of Individuals Who Refuse Participation After/During Consent Process.: The number of individuals who refuse participation after/during consent process.
Arm/Group | The Number of Individuals Who Refuse Participation After/During Consent Process.
Number analyzed (Participants) | 31
Participants | 1

6. Primary Outcome: Mean Sessions Completed
Description: The mean number of sessions completed by study participants in the MORE intervention.
Time Frame: At 8-weeks (post treatment period completion).
Population: Participants randomized to receive the MORE intervention.
Measure: Mean (Standard Deviation); unit: number of sessions
Groups:
- The Mean Number of Sessions Completed by Study Participants in the MORE Intervention.: The mean number of sessions completed by study participants in the MORE intervention.
Arm/Group | The Mean Number of Sessions Completed by Study Participants in the MORE Intervention.
Number analyzed (Participants) | 15
number of sessions | 6.4 (3.9)

7. Primary Outcome: Percentage of Sessions Completed
Description: The mean percentage of sessions completed by study participants randomized to MORE.
Time Frame: At 8-weeks (post treatment period completion).
Population: Participants randomized to MORE
Measure: Mean (Standard Deviation); unit: percentage of sessions
Groups:
- The Mean Percentage of Sessions Completed by Study Participants Randomized to MORE.: The mean percentage of sessions completed by study participants randomized to MORE.
Arm/Group | The Mean Percentage of Sessions Completed by Study Participants Randomized to MORE.
Number analyzed (Participants) | 15
percentage of sessions | 76 (.20)

8. Primary Outcome: Number Who Drop Out
Description: Number of participants who drop out of the study.
Time Frame: At 16 weeks.
Population: Participants enrolled and randomized.
Measure: Count of Participants; unit: Participants
Groups:
- Number of Participants Who Dropped Out of the Study.: Number of participants who dropped out of the study.
Arm/Group | Number of Participants Who Dropped Out of the Study.
Number analyzed (Participants) | 30
Participants | 0

9. Primary Outcome: Percentage Who Drop Out
Description: Percentage of participants who drop out of the study.
Time Frame: At 16 weeks.
Population: Participants enrolled and randomized.
Measure: Number; unit: percentage of particpants
Groups:
- Percentage of Participants Who Dropped Out of the Study.: Percentage of participants who dropped out of the study.
Arm/Group | Percentage of Participants Who Dropped Out of the Study.
Number analyzed (Participants) | 30
percentage of particpants | 0

10. Primary Outcome: Baselines Completed
Description: The number of participants who complete baseline assessments.
Time Frame: At baseline,
Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Groups:
- Baselines Completed: The number of people who completed baseline assessments.
Arm/Group | Baselines Completed
Number analyzed (Participants) | 30
Participants | 30

11. Primary Outcome: Percentage Baselines Completed
Description: Percentage of people who completed baseline assessments.
Time Frame: At baseline,
Population: All randomized participants.
Measure: Number; unit: percentage of baseline assessments
Groups:
- Percentage Baselines Completed: The percentage of people who completed baseline assessments.
Arm/Group | Percentage Baselines Completed
Number analyzed (Participants) | 30
percentage of baseline assessments | 100

12. Primary Outcome: 8-weeks Completed
Description: The number of participants who complete 8-week assessments.
Time Frame: At 8-weeks.
Population: All participants randomized.
Measure: Count of Participants; unit: Participants
Groups:
- 8-weeks Completed: The number of participants who completed 8-week assessments.
Arm/Group | 8-weeks Completed
Number analyzed (Participants) | 30
Participants | 30

13. Primary Outcome: Percentage 8-Weeks Completed
Description: Percentage of participants who completed 8-week assessments.
Time Frame: At 8-weeks.
Population: All randomized participants.
Measure: Number; unit: percentage of 8-week assessments.
Groups:
- Percentage 8-weeks Completed: The percentage of participants who completed 8-week assessments.
Arm/Group | Percentage 8-weeks Completed
Number analyzed (Participants) | 30
percentage of 8-week assessments. | 100

14. Primary Outcome: 16-Weeks Completed
Description: The number of participants who completed 16-week assessments.
Time Frame: At 16-weeks.
Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Groups:
- 16-Weeks Completed: The number of participants who completed 16-week assessments.
Arm/Group | 16-Weeks Completed
Number analyzed (Participants) | 30
Participants | 29

15. Primary Outcome: Percentage of 16-Weeks Completed
Description: Percentage of participants who completed 16-week assessments.
Time Frame: At 16-weeks.
Population: All randomized participants.
Measure: Number; unit: percentage of 16-week assessments.
Groups:
- Percentage of 16-weeks Completed: The percentage of participants who completed 16-week assessments.
Arm/Group | Percentage of 16-weeks Completed
Number analyzed (Participants) | 30
percentage of 16-week assessments. | 96.7

16. Secondary Outcome: Days of Illicit Drug Use
Description: Research staff asked participants if they used various drugs (i.e., heroin, cocaine, opioids, marijuana, amphetamines, inhalants, hallucinogens, benzodiazepines, zolpidem, methylphenidate, or other drugs) in the past 30 days and the number of days of use for each drug in the past 30 days. "Days of illicit drug use" was determined by counting the number of days each participant used drugs based on past-30 day self-reports at the16-week assessments.
Time Frame: 16-weeks
Population: All individuals randomized.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Mindfulness Oriented Recovery Enhancement | Methadone Program Behavioral Treatment as Usual
Number analyzed (Participants) | 15 | 15
days | 6.37 (2.76) | 15.56 (2.77)
Statistical Analysis 1: Comparison: Mindfulness Oriented Recovery Enhancement vs Methadone Program Behavioral Treatment as Usual; Test type: Superiority; p = .048, ANOVA

17. Secondary Outcome: Days of Illicit Opioid Use
Description: Research staff asked participants if they used illicit opioids in the past 30 days and the number of days of use for each drug in the past 30 days. "Days of illicit opioid use" was determined by counting the number of days each participant used illicit opioids based on past-30 day self-reports at the 16-week assessment.
Time Frame: 16-weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Mindfulness Oriented Recovery Enhancement | Methadone Program Behavioral Treatment as Usual
Number analyzed (Participants) | 15 | 15
days | 2.47 (.97) | 5.49 (.97)
Statistical Analysis 1: Comparison: Mindfulness Oriented Recovery Enhancement vs Methadone Program Behavioral Treatment as Usual; Test type: Superiority; p = .037, ANCOVA

18. Secondary Outcome: Opioid Craving
Description: Research staff assessed opioid craving with a version of the Penn Alcohol Craving Scale (PACS; Flannery et al., 1999) that was adapted to assess craving to opioids at 16-weeks. Scores range from 0 to 36. Higher scores indicate greater craving.
Time Frame: 16-weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Oriented Recovery Enhancement | Methadone Program Behavioral Treatment as Usual
Number analyzed (Participants) | 15 | 15
score on a scale | 15.52 (1.71) | 21.35 (1.72)
Statistical Analysis 1: Comparison: Mindfulness Oriented Recovery Enhancement vs Methadone Program Behavioral Treatment as Usual; Test type: Superiority; p = .024, ANCOVA

19. Secondary Outcome: Pain Level.
Description: Pain was assess with the pain subscale (i.e., bodily pain severity and interference) of the RAND 36-Item Short Form Health Survey. Scores range from 0 to 100, with higher scores indicating better functioning, health, and well-being and less pain, limitations, and symptom severity or interference as compared to lower scores.
Time Frame: 16-weeks
Population: All randomized participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Oriented Recovery Enhancement | Methadone Program Behavioral Treatment as Usual
Number analyzed (Participants) | 15 | 15
score on a scale | 50.76 (5.52) | 26.65 (5.54)
Statistical Analysis 1: Comparison: Mindfulness Oriented Recovery Enhancement vs Methadone Program Behavioral Treatment as Usual; Test type: Superiority; p = .005, ANCOVA

20. Secondary Outcome: Depression Level.
Description: Depression was measured with Center for Epidemiologic Studies Depression Scale (CES-D). The CES-D scale is a widely used valid and reliable measure that consists of 20 items with potential scores ranging from 0 to 60. A score above 16 on the CES-D indicates clinically significant symptoms of depression. Higher scores on the CES-D indicates greater depression.
Time Frame: 16-weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Oriented Recovery Enhancement | Methadone Program Behavioral Treatment as Usual
Number analyzed (Participants) | 15 | 15
score on a scale | 34.11 (2.31) | 42.93 (2.34)
Statistical Analysis 1: Comparison: Mindfulness Oriented Recovery Enhancement vs Methadone Program Behavioral Treatment as Usual; Test type: Superiority; p = .013, ANOVA

21. Secondary Outcome: Anxiety Level.
Description: Anxiety was measured with the Beck Anxiety Inventory (BAI). The BAI is also a widely used, reliable, and valid scale that consists of 21 items with potential scores ranging from 0 to 63. A score of 16 or higher indicates clinically sig-nificant symptoms of anxiety. A higher score on the BAI indicates greater anxiety.
Time Frame: 16-weeks
Population: All randomized participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Oriented Recovery Enhancement | Methadone Program Behavioral Treatment as Usual
Number analyzed (Participants) | 15 | 15
score on a scale | 41.05 (3.09) | 50.83 (3.09)
Statistical Analysis 1: Comparison: Mindfulness Oriented Recovery Enhancement vs Methadone Program Behavioral Treatment as Usual; Test type: Superiority; p = .035, ANOVA

ADVERSE EVENTS:
Time Frame: 16-weeks
Arm/Group | Mindfulness Oriented Recovery Enhancement | Methadone Program Behavioral Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-24): https://cdn.clinicaltrials.gov/large-docs/01/NCT03894501/Prot_SAP_000.pdf